CLINICAL TRIAL: NCT01717300
Title: A 24-Week, Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Assess the Efficacy and Tolerability of Anacetrapib When Added to Ongoing Statin Therapy With or Without Other Lipid Modifying Medication(s) in Patients With Hypercholesterolemia or Low HDL-C
Brief Title: A Study of the Safety and Efficacy of Anacetrapib (MK-0859) When Added to Ongoing Statin Therapy (MK-0859-021)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-021; 2012-003110-14 (EudraCT Number)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anacetrapib 100 mg (Experimental)
  Interventions: Drug: Anacetrapib 100 mg; Drug: Placebo for anacetrapib 25 mg
- Anacetrapib 25 mg (Experimental)
  Interventions: Drug: Placebo for anacetrapib 100 mg; Drug: Anacetrapib 25 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for anacetrapib 100 mg; Drug: Placebo for anacetrapib 25 mg

INTERVENTIONS:
Drug: Anacetrapib 100 mg — 100 mg tablet, oral, once daily for 24 weeks
  Other Names: MK-0859
  Arms: Anacetrapib 100 mg
Drug: Placebo for anacetrapib 100 mg — Placebo tablet, orally, once daily for 24 weeks
  Arms: Anacetrapib 25 mg; Placebo
Drug: Anacetrapib 25 mg — 25 mg tablet, oral, once daily for 24 weeks
  Other Names: MK-0859
  Arms: Anacetrapib 25 mg
Drug: Placebo for anacetrapib 25 mg — Placebo tablet, orally, once daily for 24 weeks
  Arms: Anacetrapib 100 mg; Placebo

SUMMARY:
This study will evaluate the effects of 2 different dose levels of anacetrapib on low-density lipoprotein-cholesterol (LDL-C) and high-density lipoprotein cholesterol (HDL-C) in participants with hypercholesterolemia when added to an existing statin-modifying therapy.

ELIGIBILITY:
Inclusion Criteria:

* If female, cannot be of reproductive potential
* Have been treated with an optimal dose of statin for at least 6 weeks
* Coronary heart disease (CHD) or other atherosclerotic vascular disease with multiple risk factors (including diabetes, metabolic syndrome) and/or high LDL-C/low HDL-C, or needing to meet a specific LDL-C/HDL-C goal

Exclusion Criteria:

* Previously participated in a study with a cholesteryl ester transfer protein (CETP) inhibitor
* Homozygous familial hypercholesterolemia
* Severe chronic heart failure
* Uncontrolled cardiac arrhythmias, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery by-pass graft (CABG), unstable angina, or stroke within 3 months
* Uncontrolled hypertension
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Active or chronic hepatobiliary, hepatic, or gall bladder disease
* History of mental instability, drug/alcohol abuse within the past five years or major psychiatric illness inadequately controlled and unstable
* History of ileal bypass, gastric bypass, or other significant condition associated with malabsorption
* Human immunodeficiency virus (HIV) positive
* History of malignancy ≤5 years
* Donated blood products or has had phlebotomy of >300 mL within 8 weeks or intends to donate 250 mL of blood products or receive blood products within the projected duration of the study
* Currently taking medications that are potent inhibitors or inducers of cytochrome P450 3A4 (CYP3A) (including but not limited to cyclosporine, systemic itraconazole or ketoconazole, erythromycin, clarithromycin, or telithromycin, nefazodone, protease inhibitors, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St John's wort) or has discontinued treatment <3 weeks prior
* Consumes more than 2 alcoholic drinks per day
* Currently participating or has participated in a study with an investigational compound or device within 3 months
* Receiving treatment with systemic corticosteroids or taking systemic anabolic agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2014-10-29 (Actual); Study Completion 2014-10-29 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in LDL-C (beta-quantification [BQ] method) | Baseline and Week 24
Percent Change from Baseline in HDL-C | Baseline and Week 24
Number of Participants with Alanine Transaminase (ALT) or Aspartate Aminotransferase (AST) Consecutive Elevations ≥3xULN (Upper Limit of Normal) | 24 Weeks
Number of Participants with Creatine Phosphokinase Elevations ≥10xULN with or without Muscle Symptoms | 24 weeks
Number of Participants with Sodium, Chloride, or Bicarbonate Elevations >ULN or Potassium Levels <LLN (Lower Limit of Normal) | 24 weeks
Number of Participants with Pre-specified Adjudicated Cardiovascular Serious Adverse Events or Death from Any Cause | 24 weeks
Number of Participants with Significant Increase in Blood Pressure | 24 weeks

SECONDARY OUTCOMES:
Percent change from Baseline in non-HDL-C | Baseline and Week 24
Percent Change from Baseline in Apolipoprotein B (Apo-B) | Baseline and Week 24
Percent Change from Baseline in Apolipoprotein A-I (Apo-A-I) | Baseline and Week 24
Percent Change from Baseline in Lipoprotein(a) (lp[a]) | Baseline and Week 24
Percent Change from Baseline in HDL-C Among Participants with Low HDL-C at LDL-C goal | Baseline and Week 24

REFERENCES:
- [Result] Ballantyne CM, Shah S, Kher U, Hunter JA, Gill GG, Cressman MD, Ashraf TB, Johnson-Levonas AO, Mitchel YB. Lipid-Modifying Efficacy and Tolerability of Anacetrapib Added to Ongoing Statin Therapy in Patients with Hypercholesterolemia or Low High-Density Lipoprotein Cholesterol. Am J Cardiol. 2017 Feb 1;119(3):388-396. doi: 10.1016/j.amjcard.2016.10.032. Epub 2016 Nov 1. PMID 27956003